CLINICAL TRIAL: NCT01084447
Title: Effect of Inspiratory Muscle Training on Muscular and Pulmonary Function Following Gastroplasty in Obese Patients
Brief Title: Inspiratory Muscle Training After Gastroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Effect of inspiratory muscle training on muscular and pulmonary function following gastroplasty in obese patients, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USP-2010
Record Dates: First submitted 2010-03-04; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Obesity
Keywords: obesity; gastroplasty; respiratory muscle training; muscle strength; physical therapy
MeSH Terms: conditions — Obesity | interventions — Breathing Exercises; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Placebo Comparator): In placebo muscular training group the respiratory exercise was used a linear pressure resistance device (Threshold ® IMT - Health Scan Products; USA) no load.
  Interventions: Device: control group
- trained group (Active Comparator): In trained group the respiratory exercise used a linear pressure resistance device (Threshold ® IMT - Health Scan Products; USA)the load was initially set at 40% of the maximal inspiratory pressure.
  Interventions: Device: inspiratory muscle training

INTERVENTIONS:
Device: inspiratory muscle training — This daily respiratory exercise was performed from the 2nd day following surgery by using a linear pressure resistance device (Threshold ® IMT - Health Scan Products; USA)was initially set at 40% of the maximal inspiratory pressure, obtained in the 2nd post-operative day, being adjusted to every new maximal inspiratory pressure measurement.
  Other Names: respiratory training
  Arms: trained group
Device: control group — In placebo muscular training the daily respiratory exercise was performed from the 2nd day following surgery by using a linear pressure resistance device (Threshold ® IMT - Health Scan Products; USA)no load until the 30th post-operative day.
  Arms: control group

SUMMARY:
The purpose of this study is to assess the effect of post-operative inspiratory muscle training on muscle strength and endurance in patients with obesity submitted to gastroplasty.

DETAILED DESCRIPTION:
Gastroplasties, like other major abdominal surgeries, induce mechanical changes in the lungs and decreases of the respiratory muscle strength in the post-operative periods. Depending on the occurrence of pre-existing disturbs, obese patients may exhibit severe declines of respiratory function after these surgeries.

Post-operative respiratory physiotherapy is a valuable intervention, involving a set of techniques aimed to expand pulmonary volumes and to improve arterial oxygenation, leading to decreases on the development of atelectasis and pneumonias. It induces faster recovery of respiratory function and reduction of lung complications, what may be particularly important in high-risk patients like over-weighted subjects.

There are scanty data about the role of respiratory muscle training in the post-operative period. This is particularly true regarding inspiratory muscle training of obese patients submitted to gastroplasties.

ELIGIBILITY:
Inclusion Criteria:

* gastroplasty patients presenting body mass index (BMI) ≥ 35 kg/m2;
* weighting ≤ 60 kg/m2;
* capable of fulfilling the experimental protocol.

Exclusion Criteria:

* acute or chronic pulmonary disease;
* smoking;
* post-operative mechanical ventilation for more than 48 hours;
* presence of lung complications;
* need for surgical re-intervention during the study period.

Ages: 20 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-01; Primary Completion 2004-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Maximum static respiratory pressures | post-operative days 2, 7, 14, and 30
  This measurement was made at mouth level by using a properly calibrated manovacuometer (GERAR ®, São Paulo, Brazil), with graduation ranging from 0 to ± 300 cmH2O, connected to a rigid plastic tube.
Inspiratory muscular endurance test | post-operative days 2, 7, 14, and 30.
  This measurement was performed by using the Threshold® IMT device (Health Scan Products, USA), at 80% maximal inspiratory pressure, in sitting position.
Spirometric measurements | post-operative days 2, 7, 14, and 30.
  Spirometry was performed according to norms of the American Thoracic Society (ATS) (1994)19 by using a previously calibrated spirometer (Respiradyne II Plus®, Sherwood Medical, St. Louis, USA).

SECONDARY OUTCOMES:
Maximum static respiratory pressures | post-operative days 2, 7, 14, and 30
Inspiratory muscular endurance test | post-operative days 2, 7, 14, and 30
Spirometric measurements | post-operative days 2, 7, 14, and 30.

CONTACTS AND LOCATIONS:
Overall Officials: Ada C Gastaldi, PHD, Principal Investigator — Faculty of Medicine of Ribeirao Preto-University of Sao Paulo
Locations (1):
- Faculty of Medicine of Ribeirão Preto, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Christensen EF, Schultz P, Jensen OV, Egebo K, Engberg M, Gron I, Juhl B. Postoperative pulmonary complications and lung function in high-risk patients: a comparison of three physiotherapy regimens after upper abdominal surgery in general anesthesia. Acta Anaesthesiol Scand. 1991 Feb;35(2):97-104. doi: 10.1111/j.1399-6576.1991.tb03255.x. PMID 2024569
- [Background] Dronkers J, Veldman A, Hoberg E, van der Waal C, van Meeteren N. Prevention of pulmonary complications after upper abdominal surgery by preoperative intensive inspiratory muscle training: a randomized controlled pilot study. Clin Rehabil. 2008 Feb;22(2):134-42. doi: 10.1177/0269215507081574. Epub 2007 Dec 5. PMID 18057088
- [Derived] Casali CC, Pereira AP, Martinez JA, de Souza HC, Gastaldi AC. Effects of inspiratory muscle training on muscular and pulmonary function after bariatric surgery in obese patients. Obes Surg. 2011 Sep;21(9):1389-94. doi: 10.1007/s11695-010-0349-y. PMID 21229331